CLINICAL TRIAL: NCT00151879
Title: A Multicenter, Open-label Trial to Investigate the Safety and Tolerability of Intravenous SPM 927 as Replacement for Oral SPM 927 in Subjects With Partial Seizures With or Without Secondary Generalization.
Brief Title: Safety and Tolerability of Intravenous SPM 927 as Replacement for Oral SPM 927 in Subjects With Partial Seizures
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0757; 2004-002322-22 (EudraCT Number)
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2010-07

CONDITIONS: Epilepsies, Partial
Keywords: partial seizures with or without secondary generalization
MeSH Terms: conditions — Epilepsies, Partial | interventions — 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-

INTERVENTIONS:
Drug: SPM 927

SUMMARY:
Subjects enrolled in the SP615, SP756, or SP774 open-label extension (OLE) trials receiving oral SPM 927 for at least 8 weeks and a stable dose of up to 3 antiepileptic medications may participate in a research trial at approximately 30 locations.

Trial objectives include investigating whether iv SPM 927 is safe and well tolerated when given twice daily for a short period of time and identifying the appropriate infusion rate(s).

Subjects will receive SPM 927 as a 30-, 15- or 10- minute infusions twice daily for 2 - 5 days based on notification by the research doctor and subject choice. Subjects will remain on the same stable dose as received in the OLE trial.

Trial procedures will include medical history update, physical/ neurological exams, ECGs, blood /urine sample collections and seizure diary completion.

Subjects completing the trial will return to the OLE trial to resume dosing with oral SPM 927.

ELIGIBILITY:
Inclusion Criteria:

* Partial seizures with or without secondary generalization.

Exclusion Criteria:

* Subject has previously received iv lacosamide.
* Subject meets the withdrawal criteria for the open-label extension trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2005-02; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of lacosamide when given as iv infusions in subjects who are receiving oral lacosamide in addition to up to 3 concomitant AEDs for partial seizures. The primary variables are adverse events

SECONDARY OUTCOMES:
Seizure counts, trough and measured maximum concentration for lacosamide as well as the O-desmethyl-metabolite.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Schwarz, RTP, North Carolina, United States

REFERENCES:
- [Result] Krauss G, Ben-Menachem E, Mameniskiene R, Vaiciene-Magistris N, Brock M, Whitesides JG, Johnson ME; SP757 Study Group. Intravenous lacosamide as short-term replacement for oral lacosamide in partial-onset seizures. Epilepsia. 2010 Jun;51(6):951-7. doi: 10.1111/j.1528-1167.2009.02463.x. Epub 2009 Dec 22. PMID 20041945